CLINICAL TRIAL: NCT03226652
Title: Heart Function in Patients Assessed for Sleep Disordered Breathing (SDB)
Brief Title: Heart Function in Patients Assessed for Sleep Apnoea
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 17IC3980
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Results first posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Sleep Disordered Breathing; Heart Failure With Normal Ejection Fraction; Obstructive Sleep Apnea; Central Sleep Apnea; Heart Failure
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Sleep Apnea, Central; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with clinically suspected sleep disordered breathing (SDB): Patients referred for Sleep disordered breathing assessment.

SUMMARY:
This study aims to determine the prevalence and prognosis of heart failure with preserved ejection function (HFpEF) among patients being assessed for sleep disordered breathing (SDB).

DETAILED DESCRIPTION:
Patients with sleep disordered breathing (SDB) and those with heart failure with preserved ejection fraction (HFpEF) share similar characteristics. Increasing age, hypertension, obesity, diabetes mellitus and atrial fibrillation are well recognised links in both groups. It also known that SDB is common in patients with heart failure, both with reduced and preserved ejection fraction. It is therefore hypothesised that among patients being referred for SDB assessment, we can identify a group with unrecognised HFpEF.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥40 years and referred for respiratory polygraphy

Exclusion Criteria:

* Previous diagnosis of Heart Failure
* Treated sleep disordered breathing

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred from primary and secondary care for SDB assessment.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin R Cowie, MD MSc, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Clinically Suspected Sleep Disordered Breathing (SDB): Patients with clinically suspected SDB investigated with respiratory polygraphy.
Period: Overall Study
Arm/Group | Patients With Clinically Suspected Sleep Disordered Breathing (SDB)
Started | 101
Completed | 101
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Clinically Suspected Sleep Disordered Breathing (SDB)
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 59
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 101

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Unrecognised Heart Failure With Preserved Ejection Fraction (HFpEF) in Cohort With Clinically Suspected Sleep Disordered Breathing (SDB)
Description: The diagnosis of HFpEF was established using criteria set out in the European Society for Cardiology (ESC) guidelines based on clinical symptoms and/or signs, biomarker analysis (NT-proBNP) and evidence of structural cardiac remodeling or diastolic dysfunction on transthoracic echocardiography.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Clinically Suspected Sleep Disordered Breathing (SDB)
Number analyzed (Participants) | 101
Participants | 7

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Patients With Clinically Suspected Sleep Disordered Breathing (SDB)
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT03226652/Prot_SAP_ICF_000.pdf